CLINICAL TRIAL: NCT00317954
Title: Spironolactone in Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2612-2233
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2005-08

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; Spironolactone; Aldosterone antagonism; Renoprotection
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
The aim of the study was to evaluate the renoprotective effect (i.e. albuminuria- and bloodpressure lowering effect) of spironolactone 25 mg o.d. in type 1 and type 2 diabetic patients with albuminuria despite recommended antihypertensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus
* Diabetic Nephropathy
* Glomerular filtration rate > 30 ml/min/1.73 m2
* Blood pressure > 130/80 mm Hg

Exclusion Criteria:

* Child bearing potential
* Plasma-potassium >4.5 mmol/l
* Breastfeeding
* Abuse of alcohol or drugs
* Non-diabetic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-09; Study Completion 2005-07

PRIMARY OUTCOMES:
Changes in albuminuria
Changes in blood pressure

SECONDARY OUTCOMES:
Changes in glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Parving, MD,DMSc,Prof, Study Chair — Steno Diabetes Center Copenhagen; Katrine J Schjoedt, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Result] Schjoedt KJ, Rossing K, Juhl TR, Boomsma F, Rossing P, Tarnow L, Parving HH. Beneficial impact of spironolactone in diabetic nephropathy. Kidney Int. 2005 Dec;68(6):2829-36. doi: 10.1111/j.1523-1755.2005.00756.x. PMID 16316360
- [Result] Rossing K, Schjoedt KJ, Smidt UM, Boomsma F, Parving HH. Beneficial effects of adding spironolactone to recommended antihypertensive treatment in diabetic nephropathy: a randomized, double-masked, cross-over study. Diabetes Care. 2005 Sep;28(9):2106-12. doi: 10.2337/diacare.28.9.2106. PMID 16123474